CLINICAL TRIAL: NCT07052136
Title: Comparison Between Efficacy of Levetiracetam Versus Valproic Acid in Pediatric Patients With Status Epilepticus
Brief Title: Efficacy Comparison Between Levetiracetam and Valproic Acid in Pediatric Patients With Status Epilepticus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DRATIFA-NISHTER
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Levetiracetam; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levetiracetam group (Experimental): In this group, patients were treated with intravenous levetiracetam (LEV) 20 mg/kg over 15 minutes, followed by 60 mg/kg/day in two divided doses over 24 hours.
  Interventions: Drug: Levetiracetam
- Valproic acid group (Experimental): Patients received intravenous valproic acid at 15 mg/kg over 15 minutes, followed by 20 mg/kg/day in two divided doses over 24 hours.
  Interventions: Drug: Valproic acid

INTERVENTIONS:
Drug: Levetiracetam — Patients were treated with intravenous levetiracetam (LEV) 20 mg/kg over 15 minutes, followed by 60 mg/kg/day in two divided doses over 24 hours.
  Arms: Levetiracetam group
Drug: Valproic acid — Patients received intravenous valproic acid at 15 mg/kg over 15 minutes, followed by 20 mg/kg/day in two divided doses over 24 hours.
  Arms: Valproic acid group

SUMMARY:
Since there is a significant degree of variability in the results of previous studies and there exists a thirst for local data regarding this topic, the current study was planned, with the objective of comparing the efficacy of levetiracetam versus valproic acid in pediatric patients with status epilepticus.

DETAILED DESCRIPTION:
Early and sustained control of seizures is paramount in status epilepticus to save the life of the patient, and this warrants the use of the best drug based on evidence. Identifying a better drug in status epilepticus would add to the local data and help clinicians in making evidence-based decisions to opt for an appropriate treatment in case of failed response to benzodiazepines.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Aged 2-14 years
* Presenting with status epilepticus

Exclusion Criteria:

* Patients with focal seizures
* Patients already using valproic acid or levetiracetam
* Patients with a history of hypersensitivity to either drug

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Sustained control of seizure activity | 24 hours
  Sustained control was labeled when there was no seizure activity on EEG and regain of consciousness for ≥ 24 hours

SECONDARY OUTCOMES:
Immediate cessation of seizure activity | 30 minutes
  Immediate cessation was defined as cessation of seizure activity within 15-30 minutes, after completion of drug infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Atifa Mazhar, Principal Investigator — Nishtar University Hospital, Multan; Javaria Rasheed, FCPS, Study Director — Nishtar University Hospital, Multan
Locations (1):
- Nishtar University Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.